CLINICAL TRIAL: NCT01761487
Title: SELECTIVE DIGESTIVE DECONTAMINATION USING ORAL GENTAMICIN AND ORAL POLYMYXIN E FOR ERADICATION OF CARBAPENEM-RESISTANT KLEBSIELLA PNEUMONIAE CARRIAGE IN HOSPITALIZED PATIENTS
Brief Title: SDD for Eradicating CRKP Carriage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0285-12
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-10

CONDITIONS: Carriers of Carbapenem-resistant Klebsiella Pneumonia

ARMS (1):
- One arm only - Gentamicin and polymyxin E (Other): All subjects will receive:Gentamicin and polymyxin E paste applied on buccal surface four times daily + gentamicin + polymyxin E PO + Strict contact precautions
  Interventions: Device: Gentamicin and polymyxin E

INTERVENTIONS:
Device: Gentamicin and polymyxin E

SUMMARY:
There is an urgent need to control the current national outbreak of Carbapenem-resistent Klebsiella pneumonia (CRKP). In Israel, the death rate among CRKP carriers is 3.5 times higher than in Carbapenem-sensitive Klebsiella pneumonia carriers (44% vs. 12.5%, respectively).

In the investigators' previous study: A Randomized, Double-Blind, Placebo-Controlled Trial of Selective Digestive Decontamination (SDD) Using Oral Gentamicin and Oral Polymyxin E for Eradication of CRKP Carriage (Infect Control Hosp Epidemiol. 2012;33:14-19) the investigators have shown that the investigators' SDD regimen is effective for decolonization patients colonized with CRKP.

The investigators' assumption is that a higher dose of polymyxin E together with gentamicin (SDD drugs) for a prolonged period is needed to overcome the likelihood of a high rate of drug inactivation in the gut, thereby reaching CRKP carriage eradication.

ELIGIBILITY:
Inclusion Criteria:

* Provide a sighed and dated written informed consent document indicating that the subject (or a legally accepted representative) has been informed of all pertinent aspects of the study
* Hospitalized men or women at least 18 years of age
* Rectal swab culture positive for CRKP in the last week
* Will be willing to initiate and remain on treatment, except for adverse events occurring

Exclusion Criteria:

* Age less than 18 years.
* Pregnant women, lactating women.
* A know allergy to one of the study drugs.
* Renal failure with creatinine clearance less than 50mL/min.
* Current Treatment with IV gentamicin and/or IV polymyxin E
* Any safety, behavioral, clinical, or administrative reasons that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
CRKP carriage at end of treatment | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Negev, Israel